CLINICAL TRIAL: NCT01444079
Title: Graft Rejection or Tolerance Affected by Serial Change of Anti-donor Lymphocyte Antibody After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0808
Record Dates: First submitted 2011-09-19; First posted 2011-09-30 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Liver Transplant Rejection
Keywords: Liver transplantation; Rejection; Tolerance
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood (serum)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver transplant recipients: Recipients who will undergo liver transplantation during study period

SUMMARY:
Liver is an organ that is well-known for its immune tolerant capacity. However, there were still controversial issues about the impact of immunologic challenge after liver transplantation on the graft function. Different results of graft function affected by immunologic factors such as pre-transplant panel reactive antibody (PRA) status, pre-transplant positive lymphocyte cross match (LCM), or post-transplant circulating donor specific antibody (DSA) has been reported according to individual institutes. There was no trial for presenting anti-donor lymphocyte antibody change after liver transplantation.

The investigators designed this study to analyze the correlation between pre- and post-transplant immune status (PRA, LCM), and graft survival / rejection episode. Also, the investigators will find aspects of anti-donor lymphocyte antibody change after liver transplantation.

DETAILED DESCRIPTION:
Study Design: Target study population is forty patients who will undergo liver transplantation for 1 year in YUHS. Pediatric and early mortality cases will be excluded. Blood sample will be collected at pre-transplant period, post-transplant 7, 14, 21 day, 3 month and 6 month.

ELIGIBILITY:
Inclusion Criteria:

* Liver recipients who undergo liver transplantation between Mar, 2011 and Feb, 2012
* Patients who can be followed for more than 3 months after transplantation

Exclusion Criteria:

* Age under 20 years
* Multi-organ transplantation
* Not agree with informed consent
* Patient who had plant to be transferred to other country or center

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult recipients who will undergo liver transplantation during study period
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
incidence of acute rejection | Time point when patients are diagnosed acute rejection
  We designed to analyze the aspects of acute rejection between anti-donor lymphocyte antibody change liver transplantation.

SECONDARY OUTCOMES:
correlation between pre- and post-transplant immune status (PRA, LCM), and graft survival | at 7 day, 14 day, 21 day after transplantation and at 3 month, 6 month after transplantation
  We designed this study to analyze the correlation between pre- and post-transplant immune status (PRA, LCM), and graft survival / rejection episode.

CONTACTS AND LOCATIONS:
Overall Officials: Myoung Soo Kim, M.D., Principal Investigator — Yonsei University College of Meidicine
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Matinlauri IH, Hockerstedt KA, Isoniemi HM. Equal overall rejection rate in pre-transplant flow-cytometric cross-match negative and positive adult recipients in liver transplantation. Clin Transplant. 2005 Oct;19(5):626-31. doi: 10.1111/j.1399-0012.2005.00364.x. PMID 16146554